CLINICAL TRIAL: NCT02397733
Title: Phase III Trial Evaluating Memory Preservation of Prophylactic Cranial Irradiation With or Without Hippocampal Avoidance in Small Cell LUNG Cancer (PREMER-TRIAL)
Brief Title: Memory Preservation of Prophylactic Cranial Irradiation With Hippocampal Avoidance (PREMER-TRIAL)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Grupo de Investigación Clínica en Oncología Radioterapia (Other)
Responsible Party: Principal Investigator, Nuria Rodriguez de Dios, Principal Investigator, Grupo de Investigación Clínica en Oncología Radioterapia
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: PREMER-TRIAL; NCT02357875 (obsolete NCT alias)
Record Dates: First submitted 2015-03-20; First posted 2015-03-25 (Estimated); Last update posted 2021-08-02 (Actual); Status verified 2021-07

CONDITIONS: Small Cell Lung Carcinoma
MeSH Terms: conditions — Small Cell Lung Carcinoma

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- Prophylactic cranial irradiation (PCI) (Active Comparator): Radiation. Prophylactic cranial irradiation : 25 Gy in 10 daily fractions, five times a week
  Interventions: Radiation: Prophylactic cranial irradiation (PCI)
- Hippocampal avoidance PCI (Experimental): Hippocampal avoidance prophylactic cranial irradiation. 25 Gy in 10 daily fractions, five times a week
  Interventions: Radiation: Hippocampal avoidance PCI

INTERVENTIONS:
Radiation: Prophylactic cranial irradiation (PCI) — Prophylactic cranial irradiation (PCI): 25 Gy in 10 daily fractions, five times a week
  Arms: Prophylactic cranial irradiation (PCI)
Radiation: Hippocampal avoidance PCI — Hippocampal avoidance prophylactic cranial irradiation 25 Gy in 10 daily fractions, five times a week
  Arms: Hippocampal avoidance PCI

SUMMARY:
The main objective of this study i sto evaluate the impact of prophylactic cranial irradiation (PCI) with hippocampal avoidance in the neurocognitive function and quality of life of small cell lung cancer patients.

In addition, the trial assesses the potential changes in hippocampal volumetry due to cranial irradiation using magnetic resonance imaging.

DETAILED DESCRIPTION:
Prophylactic cranial irradiation (PCI) has become a standard of care for selected patients with limited and extensive stage small cell lung cancer (SCLC) who have shown benefit after chemotherapy with or without thoracic radiotherapy.

Because hippocampal involvement by metastatic disease is rare, and because preclinical and clinical evidence suggests that radiation dose received by the hippocampus during whole brain radiotherapy may play a role in radiation-induced neurocognitive decline, sparing of the hippocampus during the administration of PCI should result in lower rates of memory loss.

Previous studies have demonstrated the dosimetric capabilities of intensity modulated radiation therapy (IMRT) to conformably avoid the hippocampus without detriment to the radiation dose the remaining brain receives.

The main objective of this trial is compare neurocognitive functioning following hippocampal avoidance PCI to standard PCI treatment measured by Free and Cued Selective Reminding Test (FCSRT). The FCSRT measures verbal learning and memory. The FCSRT emphasizes encoding specificity during learning and recall. One of the secondary objectives of this trial is to test the hypothesis that the lowered neurocognitive function of the patients is due to a substantial reduction in hippocampal volume in magnetic resonance imaging (MRI). Others objectives are to evaluate quality of life (QoL) and the rate of metastases in the hippocampus.

ELIGIBILITY:
Inclusion Criteria:

* New diagnosed cytological or histologically confirmed Small cell lung carcinoma (stage I-IV) candidate for PCI, for example, without progressive disease after chemo-radiotherapy in stage I-III or after response after chemotherapy in stage IV
* Performance status ≤ 1
* Negative MRI of the brain within one month before protocol entry
* Patient must give written informed consent before registration

Exclusion Criteria:

* Prior radiotherapy to the brain
* History of brain metastases
* Pregnancy or lactation

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Actual)
Dates: Start 2014-09 (Actual); Primary Completion 2019-10 (Actual); Study Completion 2020-12 (Actual)

PRIMARY OUTCOMES:
Neurocognitive functioning (NCF) (Free and Cued Selective Reminding Test) | Change from baseline to 3 months
  Free and Cued Selective Reminding Test (FCSRT) evaluated at baseline and 3 months after radiation

SECONDARY OUTCOMES:
Neurocognitive functioning (NCF) (Free and Cued Selective Reminding Test) | Change from baseline to 6,12 and 24 months
  Free and Cued Selective Reminding Test (FCSRT) evaluated at baseline and 6,12 and 24 months after radiation
Hippocampus brain metastases (brain magnetic resonance imaging) (MRI) | Change from baseline to 3, 6,12 and 24 months
  Evaluation of hippocampus brain metastases at 3, 6, 12 and 24 months after radiation
Hippocampus volume (brain magnetic resonance imaging) (MRI) | Change from baseline to 3, 6,12 and 24 months
  Evaluation of hippocampus volume at 3, 6, 12 and 24 months after radiation
Adverse effects (according to Common Toxicity Criteria for Adverse Effects) | Change from baseline to 3, 6,12 and 24 months
  Evaluation of adverse effects according to Common Toxicity Criteria for Adverse Effects (NCI-CTCAE) version 4.0 at 3, 6, 12 and 24 months after radiation
Quality of life (measured by European Organization for Research and Treatment of Cancer (EORTC) questionnaire (QLQ C-30 and QLQ BN-20) | Change from baseline to 3, 6,12 and 24 months
  Evaluation of Quality of Life (QoL) measured by European Organization for Research and Treatment of Cancer (EORTC) questionnaire (QLQ C-30 and QLQ BN-20)
Overall survival | Up to 5 years
  From the start date of PCI until the date of death from any cause, or the last follow-up date whichever came first, assessed up to 60months"

CONTACTS AND LOCATIONS:
Overall Officials: Núria Rodríguez de Dios, MD PhD, Study Chair — +34683375231
Locations (1):
- Hospital Del Mar. Radiation Oncology Department, Barcelona, Spain

REFERENCES:
- [Derived] Zeng H, Schagen SB, Hendriks LEL, Sanchez-Benavides G, Jaspers JPM, Manero RM, Lievens Y, Murcia-Mejia M, Kuenen M, Rico-Oses M, Albers EAC, Samper P, Houben R, de Ruiter MB, Dieleman EMT, Lopez-Guerra JL, De Jaeger K, Counago F, Lambrecht M, Calvo-Crespo P, Belderbos JSA, De Ruysscher DKM, Rodriguez de Dios N. Impact of HA-PCI on self-reported cognitive functioning and brain metastases in small-cell lung cancer: Pooled findings of NCT01780675 and PREMER trials. Lung Cancer. 2025 Jan;199:108036. doi: 10.1016/j.lungcan.2024.108036. Epub 2024 Nov 23. PMID 39615412
- [Derived] Ishibashi A, Kurosaki H, Miura K, Utsumi N, Sakurai H. Influence of Modulation Factor on Treatment Plan Quality and Irradiation Time in Hippocampus-Sparing Whole-Brain Radiotherapy Using Tomotherapy. Technol Cancer Res Treat. 2021 Jan-Dec;20:15330338211045497. doi: 10.1177/15330338211045497. PMID 34632876
- [Derived] Rodriguez de Dios N, Counago F, Murcia-Mejia M, Rico-Oses M, Calvo-Crespo P, Samper P, Vallejo C, Luna J, Trueba I, Sotoca A, Cigarral C, Farre N, Manero RM, Duran X, Gispert JD, Sanchez-Benavides G, Rognoni T, Torrente M, Capellades J, Jimenez M, Cabada T, Blanco M, Alonso A, Martinez-San Millan J, Escribano J, Gonzalez B, Lopez-Guerra JL. Randomized Phase III Trial of Prophylactic Cranial Irradiation With or Without Hippocampal Avoidance for Small-Cell Lung Cancer (PREMER): A GICOR-GOECP-SEOR Study. J Clin Oncol. 2021 Oct 1;39(28):3118-3127. doi: 10.1200/JCO.21.00639. Epub 2021 Aug 11. PMID 34379442
- [Derived] Rodriguez de Dios N, Counago F, Lopez JL, Calvo P, Murcia M, Rico M, Vallejo C, Luna J, Trueba I, Cigarral C, Farre N, Manero RM, Duran X, Samper P. Treatment Design and Rationale for a Randomized Trial of Prophylactic Cranial Irradiation With or Without Hippocampal Avoidance for SCLC: PREMER Trial on Behalf of the Oncologic Group for the Study of Lung Cancer/Spanish Radiation Oncology Group-Radiation Oncology Clinical Research Group. Clin Lung Cancer. 2018 Sep;19(5):e693-e697. doi: 10.1016/j.cllc.2018.05.003. Epub 2018 May 10. PMID 29891263